CLINICAL TRIAL: NCT03571958
Title: Impact of Brief Motivational Interviewing During Continuous Patient Care to Enhance Oral Hygiene
Brief Title: Brief Motivational Interviewing (BMI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DENT-2018-26921
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Motivational Interviewing, BMI, OHI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional OHI (Control) (No Intervention): Advice giving method of OHI known as "tell-show-do" to inform, demonstrate, and expect patient compliance.
- BMI (Test) (Experimental): A derivative of motivational interviewing (MI), which is a patient-centered, collaborative counseling approach to strengthen an individual's intrinsic motivation towards a positive behavior change. BMI is intended for healthcare providers with limited time (5-10 minutes) to support a positive behavior change.
  Interventions: Behavioral: BMI

INTERVENTIONS:
Behavioral: BMI — A derivative of motivational interviewing (MI), which is a patient-centered, collaborative counseling approach to strengthen an individual's intrinsic motivation towards a positive behavior change. BMI is intended for healthcare providers with limited time (5-10 minutes) to support a positive behavior change.
  Arms: BMI (Test)

SUMMARY:
The goal of this research study is to determine if the utilization of brief motivational interviewing (BMI) during continuous care is superior compared to traditional oral hygiene instruction (OHI) to reduce patients' plaque score, bleeding on probing (BOP), and gingival index (GI) longitudinal. An additional goal is to investigate chairside time of implementing BMI.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* ≥ 18 years old
* Periodontal maintenance phase (at least one year)
* Plaque score ≥30% (O'Leary plaque score)
* Minimum of two sites with BOP
* Willingness to fulfill all study requirements
* Patient of Record at the University of Minnesota School of Dentistry

Exclusion Criteria:

* Current smoker or quit smoking less than one year
* Pregnant, planning to become pregnant, or unsure of pregnancy status (self-reported)
* Uncontrolled diabetes (HbA1C > 7)
* Medical conditions that may influence the outcome of the study (neurologic or psychiatric disorders, systemic infections, cancer, and/or HIV/AIDS)
* Current use of oral bisphosphonates
* History of IV bisphosphonates
* Require pre-medication or on long-term antibiotics
* Current orthodontic treatment or planning to begin orthodontic treatment during the study
* Unable to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Plaque score | Recorded four times over a one year time frame
  Excellent hygiene: 0-20%, Good hygiene: 21-40%, Fair hygiene: 41-60%, Poor hygiene: 61-100%
Bleeding on probing (BOP) | Recorded four times over a one year time frame
  Presence of bleeding (yes) or absent of bleeding (no)
Gingival Index | Recorded four times over a one year time frame
  0= normal gingiva, 1=mild inflammation (no BOP), 2=moderate inflammation (BOP), 3=severe inflammation (spontaneous bleeding)

OTHER OUTCOMES:
Clinical attachment level | Recorded four times over a one year time frame
  Measured in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Arnett, MS, Principal Investigator — University of Minnesota
Locations (1):
- School of Dentistry, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided